CLINICAL TRIAL: NCT03983200
Title: Effect of Rotating Magnetic Therapy on Diabetic Peripheral Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Majianhua (Other)
Responsible Party: Sponsor-Investigator, Majianhua, Director, Head of Endocrinology department, Clinical Professor, Nanjing First Hospital, Nanjing Medical University
Organization: Nanjing First Hospital, Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20190530-04
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Diabetic Peripheral Neuropathy
MeSH Terms: interventions — mecobalamin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Mecobalamine 0.5mg, tid
  Interventions: Drug: Mecobalamin
- Rotating Magnetic Therapy (Experimental): Rotating Magnetic Therapy 30min,bid + Mecobalamine 0.5mg, tid
  Interventions: Device: Rotating Magnetic Therapy; Drug: Mecobalamin

INTERVENTIONS:
Device: Rotating Magnetic Therapy — Rotating Magnetic Therapy 30min, bid
  Arms: Rotating Magnetic Therapy
Drug: Mecobalamin — mecobalamine 0.5mg,tid

SUMMARY:
The aim of the study is to assess the eﬀect of Rotating Magnetic Therapy on Diabetic Peripheral Neuropathy using Nerve conduction velocity examination.

ELIGIBILITY:
Inclusion Criteria:

- 1. Volunteer to participate and sign informed consent prior to the study 2. Patients with type 2 diabetes, who met WHO1999 diagnostic criteria, had diabetes distal symmetrical multiple neuropathy (1) clear history of diabetes; (2) neuropathy at or after diagnosis of diabetes;(3) clinical manifestations and signs are consistent with DPN;(4) have clinical symptoms (pain, numbness, paresthesia, etc.), 5 examination (ankle reflex, acupuncture pain sense, vibration sense, pressure sense, temperature sense) any 1 abnormal;If there were no clinical symptoms, 2 of the 5 examinations were abnormal.(5) exclude other causes of neuropathy).

3. HbA1c<7.5%, the hypoglycemic regimen was stable for 3 months 4. No acute complications, such as diabetic ketoacidosis, diabetic hyperosmolar syndrome, etc.

Exclusion Criteria:

* 1. Patients with foreign metal bodies or pacemakers 2. Patients with a history of surgery at magnetic therapy sites within one year 3. Patients with obvious discomfort to magnetic therapy 4. Patients with bleeding or bleeding tendency 5. Patients with acute complications such as diabetic ketoacidosis 6. Impaired liver and kidney function with ALT 2.5 times higher than the upper limit of normal value;Serum creatinine was 1.3 times higher than the upper limit of normal 7. History of drug abuse and alcohol dependence in the past 5 years 8. Systemic hormone therapy was used in the last three months 9. Patients with infection and stress within 4 weeks 10. Patients who are pregnant, breast-feeding, or intending to become pregnant. 11. Any other obvious conditions or co-existing diseases determined by the researcher: such as severe cardiopulmonary diseases, endocrine diseases, neurological diseases, tumors, other pancreatic diseases, patients with a history of mental illness, or severe wasting diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-06-15 (Estimated); Primary Completion 2019-11-15 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Nerve conduction velocity examination | 1 month
  the change of Nerve conduction velocity examination

SECONDARY OUTCOMES:
MNSI | 1 month
  Michigan Neuropathy Screening Instrument
Glycosylated serum albumin | 1 month
  the change of Glycosylated serum albumin